CLINICAL TRIAL: NCT00897026
Title: ER/HER2/Ki67 Breast Cancer Subtypes as Predictive Factors for Response to Adjuvant Dose-dense Therapy, and Basal Subtypes of Double-negative Breast Cancer as Prognostic Factors in Intergroup Trial C9741
Brief Title: Studying Tissue Samples From Women Who Underwent Chemotherapy for Lymph Node-Positive Stage II or Stage IIIA Breast Cancer on Clinical Trial CLB-9741 or CLB-9344
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9741A-ICSC; U10CA031946 (NIH); CALGB-9741A-ICSC; CDR0000589237 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; In Situ Hybridization, Fluorescence; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Tissue samples are collected from patients. Tissue samples are analyzed by immunohistochemistry (Ki67, CK5/6, EGFR, ER) and fluorescence in situ hybridization (FISH).
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Genetic: fluorescence in situ hybridization; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Genetic: fluorescence in situ hybridization
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors plan the best treatment.

PURPOSE: This research study is looking at tissue samples from women who underwent chemotherapy for lymph node-positive stage II or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify biomarkers that can be used to individually tailor the use of adjuvant dose-dense therapy in women with stage II or IIIA breast cancer.

Secondary

* To identify groups of patients who have a poor prognosis despite adjuvant chemotherapy and who should be prospectively targeted for new approaches to adjuvant treatment.

OUTLINE: This is a multicenter study.

Tissue samples are collected from patients. Tissue samples are analyzed by immunohistochemistry (Ki67, CK5/6, EGFR, ER) and fluorescence in situ hybridization (FISH).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of node-positive breast cancer

  * Stage II-IIIA disease
* Underwent adjuvant chemotherapy on trial CLB-9741 or CLB-9344
* Hormone receptor status not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and older diagnosed with node-positive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2012-04-27 (Actual); Study Completion 2012-04-27 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ellis, MD, PhD, FRCP, Study Chair — Washington University Siteman Cancer Center
Locations (1):
- Washington University, St Louis, Missouri, United States